CLINICAL TRIAL: NCT04202913
Title: Building Resilience for Healthy Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-2602
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Coaching (Experimental): 1:1 Health coaching with student
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Child will receive 1:1 coaching with health coach.

SUMMARY:
School based, mental-health intervention focused on improving self-efficacy and coping skills in children aged 9-13 years. The overall premise of our intervention is that by teaching children these skills they will in-turn become more resilient when faced with life-stressors and/or adverse events.

DETAILED DESCRIPTION:
Healthy Kids is a 1:1 health coaching intervention delivered in school-settings. Students meet weekly with their assigned health coach and together they identify both strengths and areas for improvement with respect to resilience, developing resilience skills, and setting resilience goals. Topics discussed include coping skills, self-efficacy, and interpersonal relationships. The program was developed using the social determination theory (SDT), goal theory, and elements from the social-ecological model. SDT was used within the intervention to promote and facilitate behavior change. Goal theory was also utilized to develop strategies to support youth short- and long-term goal setting. Finally, weekly discussions about resilience and goal setting activities accounted for elements of the social-ecological model which acknowledges that behaviors are not independent factors, but are influenced by multiple levels of one's personal and social environment.

ELIGIBILITY:
Inclusion Criteria:

* All children in participating school

Exclusion Criteria:

* None.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 867 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Child & Youth Resilience Measure - Revised (CYRM-R) | 12 weeks
  Assessment of a child's resiliency. Scores range from 17 (low resiliency) to 85 (high resiliency)

CONTACTS AND LOCATIONS:
Overall Officials: Jill L Kaar, PhD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- Eagleview Middle School, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Unknown at this time.

REFERENCES:
- [Derived] Lee JA, Heberlein E, Pyle E, Caughlan T, Rahaman D, Sabin M, Kaar JL. Study protocol for a school-based single group pragmatic trial to promote resilience in youth: Building Resilience for Healthy Kids. Contemp Clin Trials Commun. 2021 Feb 6;21:100721. doi: 10.1016/j.conctc.2021.100721. eCollection 2021 Mar. PMID 33665468
- [Derived] Lee JA, Heberlein E, Pyle E, Caughlan T, Rahaman D, Sabin M, Kaar JL. Evaluation of a Resiliency Focused Health Coaching Intervention for Middle School Students: Building Resilience for Healthy Kids Program. Am J Health Promot. 2021 Mar;35(3):344-351. doi: 10.1177/0890117120959152. Epub 2020 Sep 22. PMID 32959670